CLINICAL TRIAL: NCT06905093
Title: Eccentric or Concentric Contralateral Training in Rehabilitation After Shoulder Surgery With Elbow Immobilization
Acronym: EXC-IMMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Sainte-Anne Military Teaching Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-CHITS-014; 2024-A02862-45 (Other: Id-RCB number)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Shoulder Surgery
Keywords: Cross-education; Contralateral training; Eccentric training; Concentric training; Immobilization; Rehabilitation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CTRL) (Active Comparator): Patients receive standard care
  Interventions: Other: Standard care
- Eccentric Training Group (EXC) (Experimental): Patients receive standard care plus eccentric training of the non-immobilized arm.
  Interventions: Other: Standard care; Other: Eccentric training of the non-immobilized arm
- Concentric Training Group (CON) (Experimental): Patients receive standard care plus concentric training of the non-immobilized arm.
  Interventions: Other: Standard care; Other: Concentric training of the non-immobilized arm

INTERVENTIONS:
Other: Standard care — Standard care including rehabilitation sessions three times per week.
Other: Eccentric training of the non-immobilized arm — The training protocol involves 3 sessions per week, separated by 24-48 hours. Each session includes 4-6 sets of 10 repetitions of elbow flexion/extension exercises on the non-immobilized arm at 60-90% of 1-RM, depending on the week. Eccentric actions are performed with controlled contraction duration (4 seconds) using a metronome. Rest periods of 2 seconds between repetitions and 2 minutes between sets are provided.
  Arms: Eccentric Training Group (EXC)
Other: Concentric training of the non-immobilized arm — The training protocol involves 3 sessions per week, separated by 24-48 hours. Each session includes 4-6 sets of 10 repetitions of elbow flexion/extension exercises on the non-immobilized arm at 60-90% of 1-RM, depending on the week. Concentric actions are performed with controlled contraction duration (4 seconds) using a metronome. Rest periods of 2 seconds between repetitions and 2 minutes between sets are provided.
  Arms: Concentric Training Group (CON)

SUMMARY:
This clinical study investigates whether contralateral training (exercising the non-immobilized arm) can help preserve muscle strength and mass in patients recovering from shoulder surgery with elbow immobilization. Immobilization is often necessary to prevent further injury, but it can lead to significant muscle loss and reduced strength, delaying recovery and increasing healthcare costs. Recent studies suggest that training the non-immobilized arm may help maintain muscle function in the immobilized arm, particularly when using eccentric exercises (where muscles lengthen under tension). This study aims to compare the effects of eccentric and concentric (shortening) contralateral training versus standard care (no training) in patients undergoing shoulder surgery.

The study involves 4 visits: pre-surgery assessments, a 4-6 weeks' immobilization period with or without training, and follow-ups at the end of immobilization, 6 weeks' post-immobilization, and 17 weeks' post-immobilization. Participants will be randomly assigned to one of three groups: a control group receiving standard care, a group performing eccentric training, or a group performing concentric training. Muscle strength, mass, and function will be measured using tests such as isometric strength, ultrasound imaging, and functional scores.

The hypothesis is that eccentric contralateral training will better preserve neuromuscular function and muscle mass in the immobilized arm compared to both standard care and concentric training. This could lead to faster recovery and improved outcomes for patients. The study will provide valuable insights into optimizing rehabilitation strategies for patients recovering from shoulder surgery.

DETAILED DESCRIPTION:
The study is structured into four visits:

* Inclusion Visit (V0): During the pre-surgical consultation, patients are informed about the study and provided with an information sheet and consent form.
* Pre-Surgery Visit (V1, PRE): Conducted within 7 days before surgery, this visit includes baseline measurements on both arms (immobilized and non-immobilized). Assessments include:

  * Isometric maximal voluntary strength of elbow flexors and extensors using an isokinetic dynamometer.
  * 1-RM (one-repetition maximum) for elbow flexors and extensors.
  * Arm circumference at 5, 10, and 15 cm from the elbow crease.
  * Anatomical cross-sectional area of arm muscles using ultrasound.
  * Forearm circumference at 5 cm from the elbow crease.
  * Handgrip strength (finger flexors).
  * Functional scores: DASH (Disabilities of the Arm, Shoulder, and Hand), Constant-Murley, joint position sense (proprioception), and muscle stiffness.
* Following surgery, patients enter a 4-6 weeks' immobilization period, during which they are randomly assigned to one of three groups:

  * Control Group (CTRL): Receives standard care, including rehabilitation sessions three times per week.
  * Eccentric Training Group (EXC): Performs standard care plus eccentric training of the non-immobilized arm.
  * Concentric Training Group (CON): Performs standard care plus concentric training of the non-immobilized arm.

The training protocol involves 3 sessions per week, separated by 24-48 hours. Each session includes 4-6 sets of 10 repetitions of elbow flexion/extension exercises on the non-immobilized arm at 60-90% of 1-RM, depending on the week. Eccentric or concentric actions are performed based on group assignment, with controlled contraction duration (4 seconds) using a metronome. Rest periods of 2 seconds between repetitions and 2 minutes between sets are provided.

• Follow-Up Visits:

* V2 (POST): At the end of immobilization, the same measurements as V1 are repeated
* V3 (POST + 6 weeks): Measurements are repeated again.
* V4 (POST + 17 weeks): Measurements are repeated again.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old) undergoing shoulder surgery (i.e., Bankart procedure, rotator cuff repair, arthroplasty)
* With an indication for immobilization, expected to last 4 to 6 weeks
* Free from any neurological pathology
* Having provided their informed consent before any participation in the research

Exclusion Criteria:

* Having a medical contraindication to the practice of physical and sports activities
* Presenting an expected modification of their physical activity of the non-immobilized limb
* Having suffered an injury to the upper limbs in the last 6 months
* Having already undergone surgery on the upper limbs
* Pregnant, parturient, and breastfeeding women
* Presenting a medically established alteration of their cognitive functions
* Subject under guardianship, curatorship, family empowerment, or judicial safeguard
* Not affiliated or beneficiary of health insurance coverage
* Any other reason that, in the investigator's opinion, could interfere with the evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Isometric maximal voluntary strength of the immobilized arm | Preoperatively and at the end of the 4-6 weeks immobilization period
  Isometric maximal voluntary strength will be assessed using an isokinetic dynamometer.

SECONDARY OUTCOMES:
Isometric maximal voluntary strength of the immobilized arm | 6 weeks and 17 weeks after immobilization
  Isometric maximal voluntary strength will be assessed using an isokinetic dynamometer.
Isometric maximal voluntary strength of the non-immobilized arm | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  Isometric maximal voluntary strength will be assessed using an isokinetic dynamometer.
Circumference of the immobilized arm and the non-immobilized arm | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  Arm circumference will be assessed in cm at 5, 10, and 15 cm from the elbow crease and forearm circumference at 5 cm from the elbow crease
Anatomical cross-sectional area of the immobilized arm and the non-immobilized arm | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  Anatomical cross-sectional area of arms muscles will be measured by ultrasound.
Maximum load, one repetition maximum (1-RM) for elbow flexors and extensors | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  Maximum load lifted once (1-RM, in kilograms) for elbow flexors and extensors of the immobilized arm and the non-immobilized arm.
Handgrip strength (finger flexors) | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  Handgrip strength in kilograms will be assessed for the immobilized arm and the non-immobilized arm.
Disabilities of the Arm, Shoulder and Hand (DASH) score | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  The DASH is a self-report 30-item questionnaire. Patients can rate difficulty and interference with daily life on a 5 point Likert scale.
  The scoring ranges from 0 for best to 100 for worst outcomes.
Constant-Murley score | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  Pain and activities of daily living are answered by the patient ; range of motion and strength are answered by the clinician.
  The possible maximum total score ranges from 0 to 100. Higher scores indicate better shoulder function.
Joint position sense (proprioception) | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  Joint position sense measurement of the immobilized arm and the non-immobilized arm.
Muscle stiffness | Preoperatively, at the end of the 4-6 weeks immobilization period, and then 6 weeks and 17 weeks after immobilization
  Muscle stiffness of the immobilized arm and the non-immobilized arm will be assessed by a device named MyotonPro. A smaller muscle stiffness indicates a better outcome.
Shoulder-SanTy Athletic Return To Sport (S-STARTS) score | 17 weeks after immobilization
  The S-STARTS test consists of 5 validated tests that assess neuromuscular control after shoulder surgery. Higher scores indicate better shoulder function.
Pain intensity of the non-immobilized arm according to a numerical rating scale (NRS) | Before and after each exercise during the 4-6 weeks immobilization period
  Pain intensity will be assessed using a Numeric Rating Scale (NRS). The minimum value of the scale, corresponding to no pain at all, is 0 and the maximum value is 10.
Borg rating of perceived exertion (RPE) scale | After each exercise during the 4-6 weeks immobilization period
  The CR-10 Borg Scale will be presented to the participants after cessation of each exercise to measure the rate of perceived exertion (RPE). Possible scores range from 0 (no effort, resting) to 10 (maximal effort).

CONTACTS AND LOCATIONS:
Overall Officials: Sergio AFONSO, Physiotherapist, Study Director — Hôpital National d'Instruction des Armées Sainte-Anne
Locations (1):
- Hôpital National d'Instruction des Armées Sainte-Anne, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No